CLINICAL TRIAL: NCT06405282
Title: The Use of Non-Invasive Imaging Devices (NIID) to Detect Temperature Differentiation and Lymphatic/Venous Flow to the Head and Neck During Head Down Tilt Position Before and After Manual Lymphatic Drainage: The NIID Study
Brief Title: Weightlessness Associated Cephalad Fluid Shifts; The Potential to Evaluate Venous and Lymphatic Dysfunction
Acronym: NIID
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Heather Barnhart, Professor, Nova Southeastern University
Other Study IDs: 2022-124
Record Dates: First submitted 2024-04-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Fluid Retention Tissue; Perfusion; Complications
Keywords: dermal flow; venous flow; fluid shift; manual lymphatic drainage; blood circulation; space simulation; diagnostic imaging; tissue temperature gradient
MeSH Terms: conditions — Edema | interventions — Manual Lymphatic Drainage; Spectroscopy, Near-Infrared; Body Temperature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy students of the Health Professions Division of NSU: Participants arrived at a predesignated room and acclimated to the ambient temperature for 15 minutes. Baseline heart rate, blood pressure, respiration rate, and oxygen saturation were taken and monitored throughout the data collection process. Participants were assessed in the HDT position (validated simulated weightlessness) for 3 hours and 45 minutes. Baseline image assessments were taken 1 minute after assuming the HDT position. Subsequent image assessments were taken every 30 minutes thereafter. Each image acquisition requires ~20 seconds and was performed by 1 of 4 trained imagers. Participants received 15 minutes of an established MLD protocol to the head, neck, and thorax before moving out of position. Immediately post-MLD, reassessment with the devices occurred. A follow-up reassessment was taken with the devices 30 minutes after MLD in the sitting position to assess potential changes and resolution of any symptoms experienced following a return to gravity environment.
  Interventions: Other: Manual Lymphatic Drainage; Device: Near infrared spectroscopy; Device: Temperature; Device: Tissue Dialectic Constant

INTERVENTIONS:
Other: Manual Lymphatic Drainage — MLD is a gentle manual technique used to decongest swollen areas and redirect lymphatic flow to non-congested areas
Device: Near infrared spectroscopy — Oxygen saturation measurement
  Other Names: Kent Snapshot
Device: Temperature — Thermal imaging
  Other Names: Long wave infrared; Wound Vision Scout
Device: Tissue Dialectic Constant — TDC captured by lymphatic fluid scanning device
  Other Names: TDC; Delfin Lymphscanner

SUMMARY:
In the weightlessness of space and significant alterations of terrestrial 1 g (1 gravity equivalent) head-to-foot hydrostatic pressure gradients, astronauts experience a dramatic fluid redistribution of ~ 2 liters from the legs to the head and neck within the first 24-48 hours of flight, among other cardiovascular and physiologic system adaptations. After only 4 days in the weightlessness of low earth orbit (LEO), changes can be seen in baroreceptor responsiveness, causing orthostatic hypotension upon subsequent return to Earth. Fluid shifts may also result in headaches, congestion or facial puffiness that can contribute to deteriorating sleep patterns. The ability to manage, mitigate, or offset these fluid shifts is vital to maintain nominal health for short and long duration space flight and potentially improve readaptation to terrestrial gravity or other surface gravity fields, such as the moon or Mars. Fluid shifts towards the cephalic region during microgravity have been speculated to contribute towards spaceflight associated neuro-ocular syndrome (SANS). SANS is a distinct, microgravity-induced phenomenon of neuro-ophthalmic findings observed in astronauts following long-duration spaceflight including choroidal folds, optic disc edema, posterior globe flattening, refractive shift, and cerebral fluid shifts noted to be persistent at 6-month post-flight MRI scans. Thus, noninvasive approaches to studying real-time fluid shifts in weightlessness could serve as critical areas of research to further SANS study and effective countermeasure protocol development. For continuous fluid shift monitoring and management, the goal is to establish baseline assessments utilizing real-time point- of-care noninvasive imaging devices (NIID).

Manual lymphatic drainage (MLD) therapy reduces lymphatic fluid in the affected limb, head, and neck to improve function and prevent progression of fluid build-up. MLD is a therapeutic massage that delivers light pressure through the skin to stimulate lymphatic vessel function. Randomized controlled trials have demonstrated statistically significant improvements in lymphatic function and pain following MLD.

The main objectives of this pilot, retrospective study were to use NIID to examine temperature differential alterations, superficial venous flow patterns (head, neck, upper torso), and venous flow patterns along the lymphatic ventromedial bundles of the medial calves and thighs when in the 6-degree head down tilt (HDT) validated space analogue position and to analyze the effect of MLD therapy administered in the HDT position on lymphatic flow and temperature. HDT is the best validated space analogue currently available for evaluation of fluid redistribution in a timely manner.

DETAILED DESCRIPTION:
Under the influence of standard developmental physiology on the Earth's surface (1 g), 70% of body fluids reside below the level of the heart. The lymphatic system has the capacity and capability to transport fluid from distal to proximal in an upward manner, against gravity and tissue pressure gradients, via lymphangion contractility, leg muscle contraction, respiratory and chest wall function, thus augmenting a "suction effect" for pumping lymphatic fluid within the subatmospheric pressure tissue distribution zones (the Guyton principle). Lymphatic drainage of the head and neck must be assisted by gravity, since these regions are above the level of the heart. In the weightlessness of space and significant alterations of terrestrial 1 g head-to-foot hydrostatic pressure gradients, astronauts experience a dramatic fluid redistribution of ~ 2 liters from the legs to the head and neck within the first 24-48 hours of flight, among other cardiovascular and physiologic system adaptations. After only 4 days in the weightlessness of LEO, changes can be seen in baroreceptor responsiveness, causing orthostatic hypotension upon subsequent return to Earth. Fluid shifts may also result in headaches, congestion, or facial puffiness that can contribute to deteriorating sleep patterns. The ability to manage, mitigate, or offset these fluid shifts is vital to maintain nominal health for short and long duration space flight and potentially improve readaptation to terrestrial gravity or other surface gravity fields, such as the moon or Mars. Fluid shifts towards the cephalic region during microgravity have been speculated to contribute towards spaceflight associated neuro-ocular syndrome (SANS). SANS is a distinct, microgravity-induced phenomenon of neuro-ophthalmic findings observed in astronauts following long-duration spaceflight including choroidal folds, optic disc edema, posterior globe flattening, refractive shift, and cerebral fluid shifts noted to be persistent at 6-month post-flight MRI scans. Thus, noninvasive approaches to studying real-time fluid shifts in weightlessness could serve as critical areas of research to further SANS study and effective countermeasure protocol development. For continuous fluid shift monitoring and management, the goal is to establish baseline assessments utilizing real-time point-of-care NIID.

MLD therapy reduces lymphatic fluid in the affected limb, head, and neck to improve function and prevent progression of fluid build-up. MLD is a therapeutic massage that delivers light pressure through the skin to stimulate lymphatic vessel function. Randomized controlled trials have demonstrated statistically significant improvements in lymphatic function and pain following MLD.

The main objectives of this pilot, retrospective case series were to use 4 standard-of-care NIIDs to examine temperature differential alterations, superficial venous flow patterns (head, neck, upper torso), and venous flow patterns along the lymphatic ventromedial bundles of the medial calves and thighs when in the 6-degree HDT space analogue position and to analyze the effect of MLD therapy administered in the HDT position on lymphatic flow and temperature. We hypothesize that dermal venous and lymphatic flow patterns of the head, neck, upper torso, and ventromedial bundle flow patterns shifted to cephalad (dermal interstitial fluid increase) and were reversed following MLD therapy in the 6-degree HDT position. More specifically, MLD therapy could alter lymphatic contractility flow patterns and interstitial fluid, in addition to temperature differentials, in the 6-degree HDT position.

The following imaging devices were used to measure fluid redistribution and temperature in the HDT: near-infrared spectroscopy imaging device (SnapShotNIR, Kent Imaging, Calgary, Canada) to capture perfusion changes through and superficial oxygenation saturation measurements; long-wave infrared and wound imaging device (WoundVision Scout, WoundVision, Indianapolis, IN) to capture thermal images measuring physiological temperature differentiation; Lymphatic fluid scanning device (LymphScanner, Delfin Technologies, Miami, FL, USA) to measure percentage water content [tissue dielectric constant (TDC)] consistent with lymphatic flow patterns and interstitial fluid alterations related to positioning.

ELIGIBILITY:
Inclusion Criteria:

* Students at Nova Southeastern University
* Aged 18-45 years
* Body Mass Index ranging from 18.5 to 24.9
* No known lymphatic dysfunction
* Written informed consent

Exclusion Criteria:

* On blood pressure medications
* On vasodilation medications
* Uses any form of nicotine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy students between the ages of 18 and 45.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Percent change (%) in TDC level from baseline | Baseline, post-30 minutes, post-60 minutes, post-90 minutes, post-120 minutes, post-150 minutes, post-180 minutes, post-195 minutes (post-MLD), and post-225 minutes (30-minutes-post-MLD)
  TDC is a measurement of local tissue water content. The lymphatic fluid scanner will assess TDC levels at the timepoints listed below. The outcome measure is the percent change in these levels to assess change in interstitial fluid in simulated microgravity; the unit is percentage.
Percent change (%) in tissue oxygenation saturation level from baseline | Baseline, post-30 minutes, post-60 minutes, post-90 minutes, post-120 minutes, post-150 minutes, post-180 minutes, post-195 minutes (post-MLD), and post-225 minutes (30-minutes-post-MLD).
  Tissue oxygenation saturation is an indicator of perfusion changes. NIRS will assess tissue oxygenation at the timepoints listed below. The outcome measure is the percent change in these levels to assess perfusion changes in simulated microgravity; the unit is percentage.
Percent change (%) in tissue temperature gradient from baseline | Baseline,post-30 minutes, post-60 minutes, post-90 minutes, post-120 minutes, post-150 minutes, post-180 minutes, post-195 minutes (post-MLD), and post-225 minutes (30-minutes-post-MLD).
  Tissue temperature gradient measures the change in temperature at an area of interest compared to surrounding tissues. Fluid shifts are associated with tissue temperature alterations. LWIT will assess the tissue temperature gradient at the timepoints listed below. The outcome measure is the percent change in temperature gradients to assess changes in thermal energy at an area of interest in simulated microgravity; the unit is percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Barnhart, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided, plan to publish summary data in peer-reviewed journal

REFERENCES:
- [Background] Michel CC. Starling: the formulation of his hypothesis of microvascular fluid exchange and its significance after 100 years. Exp Physiol. 1997 Jan;82(1):1-30. doi: 10.1113/expphysiol.1997.sp004000. No abstract available. PMID 9023503
- [Background] Debiec-Bak A, Skrzek A , Prof, Wozniewski M , Prof, Malicka I. Using Thermography in the Diagnostics of Lymphedema: Pilot Study. Lymphat Res Biol. 2020 Jun;18(3):247-253. doi: 10.1089/lrb.2019.0002. Epub 2019 Nov 19. PMID 31742482
- [Derived] Barnhart H, Aviles F Jr, Pannunzio J, Sirkis N, Hubbard C, Hardigan P, Ginsburg S, Mayrovitz H, Eckert KA, Melin MM. Using noninvasive imaging to assess manual lymphatic drainage on lymphatic/venous responses in a spaceflight analog. NPJ Microgravity. 2024 Oct 3;10(1):93. doi: 10.1038/s41526-024-00429-w. PMID 39362907